CLINICAL TRIAL: NCT03741257
Title: Hypertonic Saline 3% Compared to Hypertonic Saline 1.8% for Fluid Management of Intestinal Obstruction Surgery
Brief Title: Comparison Between Two Concentration of Hypertonic Saline in Intestinal Obstruction Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Lotfy, lecturer of anesthesia and intensive care, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N-55-2018
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Intestinal Obstruction Fluid Management With Hypertonic Saline
MeSH Terms: interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Received Hypertonic saline 3% as resuscitation fluid.
  Interventions: Drug: Hypertonic saline
- Group B (Active Comparator): Received Hypertonic saline 1.8% as resuscitation
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: Hypertonic saline — resuscitation fluid

SUMMARY:
Background and Rationale :

Perioperative fluid management is a challenging issue in surgical care especially in a procedure specific model. Recently hypertonic saline (HS) has the advantage of using the patient's own total body water by drawing interstitial space. Although it still controversial whether HS is associated with benefits in specific patient populations, particularly with respect to site of lesion and illness severity; these data provide insight into therapeutic modalities to curtail ileus formation.

Objectives :

* Measurement of total volume of fluid infused, the need of inotropic or vasopressor to maintain adequate hemodynamic parameters with assessment of electrolyte disturbances and S.lactate
* The incidence rate of surgical complications; infection and anastomotic dehiscence

Study population & Sample size :

There were no previous trials comparing the two studied groups of the current trial. We expected a small standardized effect size of 0.2. Based on this effect size, 25 subjects will be needed to elicit the difference between the two groups at an alpha level of 0.05 and power of 0.9 (Whitehead et al; 2016).

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-70 years old
* ASA≤III
* BMI 25-40kg/m.

Exclusion Criteria:

* Severe CVS diseases (EF<50%)
* Severe pulmonary diseases (Pulmonary function test ≤ 50% of predicted)
* Neurological disorders; Psychological diseases, demyelinating lesions, Parkinsonism, motor or sensory disorders.
* Pregnancy.
* Severe chronic renal disease (s. Creatinine> 2gm/dl or patients on dialysis).
* Severe hepatic impairment (Child & Pugh classification class C).
* Acid-base and electrolytes disturbances.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Total volume of infused fluids | 24 hours
  the total volume of fluids given to subjects intraoperatively and postoperatively

SECONDARY OUTCOMES:
surgical complications rate | 4 days
  the rate of surgical complications i.e leakage and wound dehisence

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes